CLINICAL TRIAL: NCT05075707
Title: Magnetic Field and Laser Therapy in Management of Diabetic Trigeminal Neuralgia
Brief Title: Comparison Between Magnetic Field and Laser Therapy in Management of Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Amira Hussin Hussin Mohammed, Assistant. Professor of physical therapy, Department of Physical Therapy for Pediatrics, Delta University for Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: magnetic and laser therapy
Record Dates: First submitted 2021-09-19; First posted 2021-10-13 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Magnetic Field Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Participants will receive the descriptive medication by neurologist
- electromagnetic group (Experimental): Participants will receive the descriptive medication by neurologist in addition to electromagnetic therapy. Electromagnetic therapy will be applied for 20 min/session for three days each week for two months.
  Interventions: Other: Electromagnetic therapy.
- low laser therapy group (Experimental): Participants will receive the descriptive medication by neurologist in addition to low laser therapy. Low laser therapy will be applied for 20 min/session for three days each week for two months.
  Interventions: Other: Low level laser therapy (LLLT)

INTERVENTIONS:
Other: Electromagnetic therapy. — Electromagnetic therapy will be applied for 20 min/ session for (3 days/ week for two months) to the group intervention.
  Arms: electromagnetic group
Other: Low level laser therapy (LLLT) — Low level laser therapy (LLLT) will be applied for 20 min/session laser scanner for three days each week for two months to the group intervention.
  Arms: low laser therapy group

SUMMARY:
Trigeminal neuralgia (TN) was defined by The International Association for the Study of Pain (IASP) as severe, sudden, usually unilateral, stabbing, brief, recurrent attacks of pain in one or more distributional branches of the trigeminal nerve. The purpose of the current study will to investigate the effect of Low level laser therapy versus electromagnetic therapy on diabetic trigeminal neuralgia pain intensity and amplitude of the compound muscle action potential of the masseter and temporalis muscles in diabetic TN patients.

ELIGIBILITY:
Inclusion Criteria:

* All participants will between the ages of 25 and 45, will of both sexes (male and female), diabetic type two patients with chronic trigeminal neuralgia, (from three to six months).
* Patients will awake, cooperative, and free of psychiatric issues (as determined by a psychologist) as well as difficulties resulting from orthopaedic or special sensory deficits.

Exclusion Criteria:

* Patients will ruled out if they developed TN due to a tumour, herpes zoster, or any other reason other than diabetes, such as significant coagulation dysfunction, cardiopulmonary dysfunction or previous invasive treatment (ethanol, radiofrequency, Gama-knife microvascular decompression, glycerinum injection).
* They will not have a previous disability in the face.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-02-22 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Studies using electromyography and complex muscle action potentials | at the beginning of the study
  All patients' compound motor action potential amplitudes in the masseter and temporalis muscles will be evaluated before interventions.
Studies using electromyography and complex muscle action potentials | by the end of successful two month of intervention
  All patients' compound motor action potential amplitudes in the masseter and temporalis muscles will be evaluated after two month of interventions.
Visual analogue scale (VAS) | at the beginning of the study
  All the participants were instructed to express their pain by Visual analogue scale (VAS) before the interventions.
Visual analogue scale (VAS) | by the end of successful two month of intervention
  All the participants were instructed to express their pain by Visual analogue scale (VAS) after two month of interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- AAA, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available to other researchers after 12 month from publishing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After 12 month from publishing.